CLINICAL TRIAL: NCT05097495
Title: The Effect of the Use of Non-Nutritive Sucking vs Non-Nutritive Sucking Combined With Breast Milk on the Neonatal Comfort During Diaper Change in Preterm Infants
Brief Title: Non-Nutritive Sucking vs Non-Nutritive Sucking Combined With Breast Milk on the Neonatal Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Zehra Kan Onturk, Assist. Prof., Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATADEK-2021/15
Record Dates: First submitted 2021-10-11; First posted 2021-10-28 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Infant, Premature
Keywords: Non Nutritive Sucking; Preterm Infant; Comfort
MeSH Terms: conditions — Premature Birth | interventions — Milk, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Only NNS) (Experimental): NNS will be started 5 minutes before diaper change. The use of NNS will continue during diaper change and up to 5 minutes after the application.
  Interventions: Procedure: Only NNS
- Experimental Group (NNS Combined with Breast Milk) (Experimental): NNS combined with breast milk will be started 5 minutes before diaper change. The use of NNS combined with breast milk will continue during diaper change and up to 5 minutes after the application.
  Interventions: Procedure: NNS Combined with Breast Milk

INTERVENTIONS:
Procedure: Only NNS — Before the procedure, the Premature Infant Comfort Scale shall be filled out.
  Procedure steps for the control group:
  * Materials shall be prepared (napkins, non-sterile gloves, pacifier)
  * Hands shall be washed; gloves shall be worn.
  * The infant shall be given a NNS just before the procedure and continue until the 5th minute after the procedure.
  * The diapers shall be changed.
  * Hands shall be washed after the procedure.
  * The Premature Infant Comfort Scale shall be assessed during, shortly after, and 5 minutes after the procedure.
  Arms: Control group (Only NNS)
Procedure: NNS Combined with Breast Milk — * Before the procedure, the Premature Infant Comfort Scale shall be filled out.
  * Materials shall be prepared (napkins, non-sterile gloves, pacifier, breast milk, cup)
  * Hands shall be washed; gloves shall be worn.
  * The cylindrical part of a pacifier shall be in touch with breast milk for 5 seconds. The infant shall be given the pacifier, combined with breast milk, just before the procedure and continue until the 5th minute after the procedure.
  * The diapers shall be changed.
  * Hands shall be washed after the procedure.
  * The Premature Infant Comfort Scale shall be assessed during, shortly after, and 5 minutes after the procedure.
  Arms: Experimental Group (NNS Combined with Breast Milk)

SUMMARY:
The aim of the study is to determine the effect of the use of non-nutritive sucking vs non-nutritive sucking combined with breast milk on neonatal comfort during diaper change in preterm infants.

DETAILED DESCRIPTION:
Newborns are faced with many painful interventions including tactile stimulation such as diaper change, axillary temperature measurement, intraoral and endotracheal aspiration during the postnatal period in the Neonatal Intensive Care Units (NICU) at the beginning of their lives. Painful interventions negatively affect the physiological parameters, comfort, sleep, growth and hospital stay of newborns. As a result of these interventions, the stress level increases in preterm infants. Increased stress level can cause long-term sequelae, risk of intraventricular hemorrhage, increased oxygen consumption and hypertension. In addition, the increased stress experience may make the infant sensitive to pain and stress in other periods of his life.

This randomized controlled prospective study was planned to be conducted in the NICU of a private hospital with branches in Istanbul until the whole sample group would be reached.

In the NICU, where the study will be conducted, preterm infants will be divided into two groups as control and experimental groups. Non-nutritive sucking (NNS) combined with breast milk will be used during diaper change for newborns in the experimental group, and only NNS will be used in the control group. NNS will be given to both groups 5 minutes before diaper change. The comfort level of the newborns will be measured with the Premature Infant Comfort Scale before the NNS, 5 minutes after the NNS, during the procedure, immediately after the procedure and 5 minutes after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* The preterm infants whose parents agree to participate in the research and sign the informed consent form;
* Who have no congenital anomaly;
* Who have no chronic disease;
* Who have undergone no surgical procedure;
* Who have no neurological symptoms;
* Who have no NEC (necrotizing enterocolitis) diagnosis;
* Who are not sedated;
* Who are not hypoglycemic;
* Who have been administered no pharmacological analgesic method 4 hours before;
* Who are born between ≥28 and ≤36+6 gestation weeks, or are in between ≥28 and ≤36+6 gestation weeks during the procedure.

Exclusion Criteria:

* The infants whose parents do not agree to participate in the research and do not sign the informed consent form;
* Who have a congenital anomaly;
* Who have a chronic disease;
* Who had undergone a surgical procedure;
* Who have neurological symptoms;
* Who have NEC (necrotizing enterocolitis) diagnosis;
* Who are sedated;
* Who are hypoglycemic;
* Who have been administered no pharmacological analgesic method 4 hours prior;
* Who were between <28 and >36+6 gestation weeks.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Change in Comfort Level | 5 minutes before, immediately before, during, immediately after, and 5 minutes after the procedure.The change in these time intervals will be assessed.
  Infant's comfort level is evaluated with Premature Infant Comfort Scale.Premature Infant Comfort Scale (PICS), which is a multidimensional scale used in evaluating comfort and pain behaviorally and psychologically. The lowest score obtained from the scale is 35, and the highest score is 7. A high score on the scale indicates a low level of comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Kan Öntürk, Assist Prof, Principal Investigator — Acibadem University
Locations (1):
- Şişli Kolan International Hastanesi, Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibbins S, Stevens B. Mechanisms of sucrose and non-nutritive sucking in procedural pain management in infants. Pain Res Manag. 2001 Spring;6(1):21-8. doi: 10.1155/2001/376819. PMID 11854758
- [Result] Lyngstad LT, Tandberg BS, Storm H, Ekeberg BL, Moen A. Does skin-to-skin contact reduce stress during diaper change in preterm infants? Early Hum Dev. 2014 Apr;90(4):169-72. doi: 10.1016/j.earlhumdev.2014.01.011. Epub 2014 Feb 16. PMID 24548816
- [Result] De Bernardo G, Riccitelli M, Sordino D, Giordano M, Piccolo S, Buonocore G, Perrone S. Oral 24% sucrose associated with nonnutritive sucking for pain control in healthy term newborns receiving venipuncture beyond the first week of life. J Pain Res. 2019 Jan 8;12:299-305. doi: 10.2147/JPR.S184504. eCollection 2019. PMID 30662283
- [Result] Naughton KA. The combined use of sucrose and nonnutritive sucking for procedural pain in both term and preterm neonates: an integrative review of the literature. Adv Neonatal Care. 2013 Feb;13(1):9-19; quiz 20-1. doi: 10.1097/ANC.0b013e31827ed9d3. PMID 23360853
- [Result] Wu HP, Yang L, Lan HY, Peng HF, Chang YC, Jeng MJ, Liaw JJ. Effects of Combined Use of Mother's Breast Milk, Heartbeat Sounds, and Non-Nutritive Sucking on Preterm Infants' Behavioral Stress During Venipuncture: A Randomized Controlled Trial. J Nurs Scholarsh. 2020 Sep;52(5):467-475. doi: 10.1111/jnu.12571. Epub 2020 Jun 20. PMID 32564489